CLINICAL TRIAL: NCT04739163
Title: Translation and Cross-cultural Adaptation of the Duke Activity Status Index to Urdu
Brief Title: Urdu Translation of Duke Activity Status
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00783 Abdul Majid Saeed
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Heart Diseases
Keywords: Duke activity status index; Heart Diseases; Tool Translation
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To translate, culturally adapt, and validate the Duke Activity Status Index (DASI) to the Pakistani Urdu language. The study will measure the reliability & validity of DASI in the Urdu version.No study has been conducted in the Pakistan region to translate DASI which follows the proper cross-culture adaptation.

DETAILED DESCRIPTION:
Literature suggested that Duke Activity Index (DASI) is a questionnaire originally developed in English To evaluate the functionality. DASI was used primarily to assess patients with cardiovascular diseases such as coronary artery disease, heart failure, myocardial ischemia, and infarction. In clinical practice, DASI can be used to know the effects of medical treatments and cardiac rehabilitation and to assist clinical decisions In controlled clinical trials, DASI can also be used to assess interventions and as a component for assessing the costs/benefits of treatment.

Studies demonstrated that DASI is characterized as a questionnaire with good functional ability, evidence of validity, usefulness, and great clinical and scientific applicability, it seems to be a useful tool for evaluating cardiac patients. So, to be used with Brazilian CVD patients it is necessary to validate DASI and verify its psychometric properties in this population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals have enough education level to understand Urdu and English as well with a body mass index between 18.6 and 39.9 kg/m with the diagnosis of cardiovascular diseases such as coronary artery disease, valvular heart disease, arrhythmia with at least one symptom11 such as chest pain, palpitations, fatigue, or dyspnea, and physician referral to exercise testing.

Exclusion Criteria:

* Individual is unable to read the questionnaire, who have cognitive deficits screened by Mini-Mental State Examination according to the cut-off points and Hospitalization two months before as well as acute illness, fever, or severe physical limitation that would prevent from doing the exercise test.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: To meet inclusion criteria participants will be diagnosed with heart disease, clinically stable, and able to read the Urdu version of DASI. Then patient response will be checked on the translated Urdu version.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Translation of Duke Activity Status Index (DASI) in Urdu | 6 months
  The Duke Activity Status Index Scale (DASI) is a questionnaire, originally developed in English to assess the functional capacity. DASI has been used mainly to evaluate patients with cardiovascular diseases, such as coronary artery disease, heart failure, myocardial ischemia and infarction.

SECONDARY OUTCOMES:
validity & reliability of Duke Activity Status Index Scale (DASI) in Urdu version | 6 months
  Reliability and validity are concepts used to evaluate the quality of research. They indicate how well a method, technique or test measures something. Reliability is about the consistency of a measure, and validity is about the accuracy of a measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- AllamaIqbal hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung SC, Hlatky MA, Stone RA, Rana JS, Escobedo J, Rogers WJ, Bromberger JT, Kelsey SF, Brooks MM. Body mass index and health status in the Bypass Angioplasty Revascularization Investigation 2 Diabetes Trial (BARI 2D). Am Heart J. 2011 Jul;162(1):184-92.e3. doi: 10.1016/j.ahj.2011.03.019. PMID 21742107
- [Background] Scotto CJ, Waechter DJ, Rosneck J. Adherence to prescribed exercise and diet regimens two months post-cardiac rehabilitation. Can J Cardiovasc Nurs. 2011;21(4):11-7. PMID 22165501
- [Background] George MJ, Kasbekar SA, Bhagawati D, Hall M, Buscombe JR. The value of the Duke Activity Status Index (DASI) in predicting ischaemia in myocardial perfusion scintigraphy - a prospective study. Nucl Med Rev Cent East Eur. 2010;13(2):59-63. PMID 21598228
- [Background] Coutinho-Myrrha MA, Dias RC, Fernandes AA, Araujo CG, Hlatky MA, Pereira DG, Britto RR. Duke Activity Status Index for cardiovascular diseases: validation of the Portuguese translation. Arq Bras Cardiol. 2014 Apr;102(4):383-90. doi: 10.5935/abc.20140031. Epub 2014 Feb 17. PMID 24652056